CLINICAL TRIAL: NCT01661660
Title: Ecological Assessment of Autonomy and Apathy in Alzheimer Patients at Mild and Moderate Stages, as Welle as in Healthy Control Particpants
Brief Title: Ecological Assessment of Autonomy and Apathy
Acronym: Dem@Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 12-PP-01
Record Dates: First submitted 2012-07-06; First posted 2012-08-09 (Estimated); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Predemential Alzheimer Patient; Demential Alzheimer Patient; Witness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control subjects (Active Comparator): Control subjects were people with memory complaints coming for a consultation and prevention.
  Interventions: Other: observationnal
- Predementia / MCI patients (Experimental): Subjects at predementia stage or MCI stage
  Interventions: Other: observationnal
- Dementia patient (Experimental): Subjects at demential stage
  Interventions: Other: observationnal

INTERVENTIONS:
Other: observationnal — Observation during a physical exercise

SUMMARY:
Cognitive symptoms are the core feature of Alzheimer's disease. Besides these problems, behavioural and psychological symptoms (BPSD), and an impairment of activities of daily living (IADL) are frequently encountered and usually show an impact on autonomy maintenance, prognostic and care during the prodromal and early stages of the disease.

Such symptoms are noticeable before the diagnosis of dementia and their occurrences as well as their intensity increase with the evolution of the disease.

Apathy, initially defined as a reduction of motivated behaviours, is the most frequently observed BPSD. Apathy is clinically defined by a significant reduction or complete loss of interest, initiative capacity and emotional blunting. Accordingly, apathy is characterized by diminished goal-directed cognitions and behaviours.

Behavioural and psychological assessment relies essentially on neuropsychiatric scales. These are used to gather precise data regarding patient's clinical state from interviews with the patient, the career or from clinical impressions during the consultation. From their apparent simplicity they have made their way into daily clinical practices, yet neuropsychiatric scales are reportedly biased by the assessors' subjectivity.

However, some tools whose allow simple, fast and objectively valid assessments are not widely used.

Hence, the use of ICT such as actigraphy (wearable device assessing locomotion activities), automatized audio-video recognition and signal analysis from events, may be of interest in addition to current assessment methods.

The aim of this study is to implement an objective assessment of goal directed activities and autonomy in an experimental design including predefined actions. The setting includes video cameras, microphones, actigraphic and Galvanic Skin Response sensors for recording and computer-based recognition of events using audio-video data, locomotion data and sinusal variability respectively as well as extracting biomarkers for supporting detection of dementia at early stages and supporting ongoing tracking of the dementia disease state. The following population will be included: patients with Mild Cognitive Impairment (n=50), patients with Alzheimer's disease (n=50) and control participants (n=50).

This work will provide further objective information for clinical practitioner in order to detect behavioral disturbances such as apathy.

ELIGIBILITY:
Subjects control Inclusion criteria

* Male or Female ≥ 65 years
* Subjects were not accompanied by an Alzheimer subject recruited for the study;
* Subjects showing no locomotor disability;
* Subjects with no cognitive impairment overall with a score> 27 on the MMSE.

Special cases:

people with no schooling aged 50 to 79 years we take a MMSE> 22/30 and for over 80 years a MMSE> 21/30 - by the standards of Kalafat, 2003) (Folstein, Folstein et al. 1975), or arguments in favor of the following diagnosis: probable Alzheimer's disease according to the criteria of the NINCDS-ADRDA and / or major depressive episode according to DSM-IV-R;

* Subjects receiving a social security system;
* Signature of informed consent.

Exclusion Criteria

* Failure to perform the protocol due to a mobility impairment;
* Prescription of a new psychotropic medication (hypnotic, anxiolytic, antidepressant, antipsychotic) in the week preceding the assessment;
* Patients implanted with a pacemaker;
* Patient Trust under curatorship or judicial protection;
* Detainees (administrative or judicial).

Predementia / MCI Patients Inclusion criteria

* Men or women ≥ 65 years.
* Subjects with a diagnosis of MCI according to the criteria of the National Institute on Ageing and Alzheimer's Association group (Albert MS, 2011, see Appendix B), or Alzheimer's disease stage prédementiel (B. Dubois, 2010; see Appendix C)
* Subjects with a score of 0 to items of "tremors" and "muscle stiffness" of the UPDRS III
* Subjects with no criteria for major depressive episode according to DSM IV-R;
* Subjects receiving a social security system;
* Signature of informed consent. Exclusion Criteria
* Failure to pass neuropsychological testing because of a sensory or motor deficit;
* Prescription of a new psychotropic medication (hypnotic, anxiolytic, antidepressant, antipsychotic) in the week preceding the assessment;
* Patients implanted with a pacemaker;
* Patient Trust under curatorship or judicial protection.

dementia subjects Inclusion criteria

* Men and women older than 65 years
* Subjects with a diagnosis of Alzheimer's disease according to NINCDS-ADRDA (McKhann, Drachman et al. 1984) or Alzheimer's typical or atypical (B. Dubois et al. 2007)
* MMSE score ≥ 16
* Subjects with a score of 0 to items of "tremors" and "muscle stiffness" of the UPDRS III
* Subjects with no criteria for major depressive episode according to DSM IV-R;
* Subjects receiving drug treatment by acetylcholinesterase inhibitor or memantine in standard dose and stable for at least 3 months;
* Subjects receiving a social security system;
* Signature of informed consent.

Exclusion Criteria

* Failure to pass neuropsychological testing because of a sensory or motor deficit;
* Prescription of psychotropic medication (hypnotic, anxiolytic, antidepressant, antipsychotic) in the week preceding the assessment;
* Patients implanted with a pacemaker
* Patient Trust under curatorship or judicial protection.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 126 (Actual)
Dates: Start 2012-06-25 (Actual); Primary Completion 2015-12-01 (Actual); Study Completion 2015-12-01 (Actual)

PRIMARY OUTCOMES:
the evaluation score of autonomy | It will be evaluated at time = 0 for each patient
  The primary outcome used to differentiate patients with Alzheimer's disease in pre-demented control subjects is the evaluation score of autonomy calculated from data collected during the execution of step semi directed

SECONDARY OUTCOMES:
analyze differences between inter-group patients | It will be evaluated at time = 0 for each patient
  The impact of behavioral problems in activities of daily living will be evaluated using the same criteria for evaluating the main objective analysis by an international group in a category between subjects diagnosed patients apathetic and not apathetic. Actigraphy data, recorded from the ecological assessment in experiment room until the end of the final medical examination, will quantify and qualify the motor activity of the subject at its presence on the premises of CMRR to compare these measures during the evaluation phases in experiment room, consulting and outside these two periods.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe ROBERT, PU-PH, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- CHU de Nice- Hôpital Cimiez_ CMRR, Nice, France